CLINICAL TRIAL: NCT07139054
Title: 68Ga-Labeled Fibroblast Activation Protein Inhibitor PET/CT for the Prediction of Clinical Response to Neoadjuvant Therapy in Nasopharyngeal Carcinoma Patients: A Prospective Study
Brief Title: 68Ga-FAPI-46 PET/CT for the Prediction of Clinical Response to Neoadjuvant Therapy in Nasopharyngeal Carcinoma Patients
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Other Study IDs: XMFHIIT-2025SL118
Record Dates: First submitted 2025-08-10; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Nasopharyngeal Cancer
MeSH Terms: conditions — Nasopharyngeal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The goal of this clinical trial is to learn about the prediction of clinical response to neoadjuvant therapy in nasopharyngeal carcinoma patients via 68Ga-FAPI-46 PET/CT. The main question it aims to answer is:

Can 68Ga-FAPI-46 PET/CT be used to evaluate the therapeutic response of neoadjuvant therapy for nasopharyngeal carcinoma？ The researchers will compare the correlation between the parameters obtained after three 68Ga-FAPI-46 PET/CT scans and the treatment response after neoadjuvant and neoadjuvant combined with concurrent chemoradiotherapy.

Participants will:

Undergo three 68Ga-FAPI-46 PET/CT scans before starting treatment, after neoadjuvant therapy, and after concurrent chemoradiotherapy

ELIGIBILITY:
Inclusion Criteria:

* Individuals of either gender, aged between 18 and 70 years;

  * Histopathologically confirmed non-keratinizing nasopharyngeal carcinoma (WHO type II or III);

    * Clinical stage III-IVa according to the AJCC/UICC 8th edition criteria, with no evidence of distant metastasis;

      * ECOG performance status score of 0 or 1;

        * No prior anti-tumor treatment, including radiotherapy, chemotherapy, immunotherapy, or biological therapy, for nasopharyngeal carcinoma; ⑹ No contraindications to radiotherapy or chemotherapy; ⑺ Adequate major organ function as defined by the following criteria:

          1. Hematologic criteria: WBC ≥ 4.0 × 10⁹/L, ANC ≥ 1.5 × 10⁹/L, PLT ≥ 100 × 10⁹/L, HGB ≥ 90 g/L (without blood transfusion, blood products, or hematopoietic growth factors such as G-CSF within the past 14 days);
          2. Biochemical criteria: ALT and AST ≤ 2.5 × upper limit of normal (ULN); BUN and CRE ≤ 1.5 × ULN or creatinine clearance ≥ 60 ml/min (calculated using the Cockcroft-Gault formula); ⑻ Willing participation in the study, with signed informed consent, good compliance, and willingness to cooperate with follow-up procedures.

             Exclusion Criteria:

          <!-- -->

          1. The pathological type was keratinizing squamous cell carcinoma or basal-like squamous cell carcinoma.
          2. Patients with a history of prior or concurrent malignant tumors that have not been cured, excluding cured basal cell carcinoma of the skin, cervical carcinoma in situ, and superficial bladder cancer;
          3. Participation in other clinical trials;
          4. Pregnant or lactating women;
          5. Uncontrolled cardiovascular diseases, including myocardial ischemia or myocardial infarction of Grade II or higher, poorly controlled arrhythmias (including a QTc interval ≥ 470 ms); patients with NYHA Class III-IV heart failure or left ventricular ejection fraction (LVEF) < 50% as assessed by echocardiography; myocardial infarction within the past year;
          6. Other severe comorbidities such as uncontrolled hypertension, severe cerebrovascular disease, severe renal disease, uncontrolled diabetes mellitus, and other chronic debilitating conditions;
          7. A history of substance abuse or alcohol dependence, psychiatric disorders, or individuals with no or limited civil capacity;
          8. According to the investigator's judgment, the subject has familial or social factors that may lead to premature termination of participation in the study, potentially affecting the subject's safety or the integrity of the study data;
          9. Patients with known hypersensitivity to ethanol.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced nasopharyngeal carcinoma in the First Affiliated Hospital of Xiamen University.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-08-10 (Actual)

PRIMARY OUTCOMES:
Treatment response to neoadjuvant therapy in patients with nasopharyngeal carcinoma | Baseline, after induction chemotherapy and before concurrent chemoradiotherapy, after concurrent chemoradiotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, China